CLINICAL TRIAL: NCT02307032
Title: Atrial Fibrillation Prediction Trial of the Dynamic Changes Through the Continuous Spectrum of the Arrhythmia Evolution.
Brief Title: Atrial Fibrillation Prediction Trial.
Acronym: AFPRET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, PETROS ARSENOS, Petros Arsenos, MD, PhD, University of Athens
Other Study IDs: 3037SH; 07062011 (Other: Sismanogleion Hospital Marousi Greece)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation Relapses Prediction; P wave Signal Averaged ECG; P wave Wavelets; Strain; Tissue Doppler Imaging
MeSH Terms: conditions — Atrial Fibrillation; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Atrial Fibrillation (AF) is a common arrhythmia with a prevalence of 1.5-2%. This prevalence increases significantly after 80 years of age. After the appearance of first episode(s) some of the patients will present frequent arrhythmia recurrences moving from the paroxysmal status to the persistent and the permanent status of the continuous spectrum of the natural time course of AF. In contrast some other will not present further relapses. To study and predict the dynamic evolution of AF is clinically important, furthermore, the detection of different sub populations risk for AF relapses will determine and different therapeutic approaches.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is a common arrhythmia with a prevalence of 1.5-2%. This prevalence increases significantly after 80 years of age. In the presence of the Arrhythmia the risk of stroke increases five fold while the congestive heart failure and the mortality rates are increasing significantly also.After the appearance of first episode(s) some of the patients will present frequent arrhythmia recurrences moving from the paroxysmal status to the persistent and the permanent status of the continuous spectrum of the natural time course of AF. In contrast some other will not present further relapses. To study and predict the dynamic evolution of AF is clinically important, furthermore, the detection of different sub populations risk for AF relapses will determine and different therapeutic approaches. The study will include > 500 patients 30-80 years old. Inclusion criteria is one up to five paroxysmal AF (PAF) episodes during the last three years. Patients during screening must maintaining Sinus Rhythm. Exclusion criteria are substrate of severe valvular diseases, congenital heart disease, previous heart surgery, hyperthyroidism, severe diseases of the autonomic nervous system, alcoholism, diseases affecting seriously the survival and absence of adequate cooperation for the study. Screening will include 12 lead surface digital ECG, 30 min High Resolution (1000 Hz) ECG recording from 3 pseudo orthogonal x,y,z leads system, and complete ECHO study (2D, PWD, TDI, Strain).Among other indices will be analyzed: P duration, P index, P dispersion, P wave signal for Late potentials, for Wavelets, PQ/RR Dynamics, Heart Rate Dynamics and various markers for the autonomic nervous system status.Primary end point is one or more PAF relapse(s) during a period of 12 months after recruitment in study.Secondary end point is permanent AF during a period of 36 months after recruitment in study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria is one up to five paroxysmal AF (PAF) episodes during the last three years. Patients during screening must maintaining Sinus Rhythm.

Exclusion Criteria:

* previous heart surgery, hyperthyroidism, severe diseases of the autonomic nervous system, alcoholism, diseases affecting seriously the survival and absence of adequate cooperation for the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include > 500 patients 30-80 years old.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation Relapse | 12 months
  Primary end point is one or more PAF relapse(s) during a period of 12 months after recruitment in study.

SECONDARY OUTCOMES:
Permanent Atrial Fibrillation | 36 months
  Secondary end point is permanent AF during a period of 36 months after recruitment in study.

CONTACTS AND LOCATIONS:
Overall Officials: Petros Arsenos, MD, PhD, Principal Investigator — First Department of Cardiology, Medical School, National & Kapodistrian University of Athens, Greece
Locations (4):
- Greece (4):
  - Cardiology Department, Hippokration Hospital, Athens, Attica
  - First Department of Cardiology, Medical School, National & Kapodistrian University of Athens, Athens, Attica
  - Cardiology Department Thriasio Hospital, Eleysina, Attica
  - Cardiology Department, Sismanogleion Hospital, Marousi